CLINICAL TRIAL: NCT05574894
Title: Effect of GH Supplementation on the Blastocyst Euploid Rate in AMA Patients--A Retrospective Cohort Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIAI E2022-022
Record Dates: First submitted 2022-10-03; First posted 2022-10-12 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-10

CONDITIONS: Growth Hormone; Advanced Maternal Age; PGT-A
MeSH Terms: interventions — Growth Hormone; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GH group (Experimental): Growth Hormone supplement, GnRH antagonist protocol for ovarian stimulation
  Interventions: Drug: Growth hormone; Drug: GnRH antagonist
- Control group (Active Comparator): No Growth Hormone supplement, GnRH antagonist protocol for ovarian stimulation
  Interventions: Drug: GnRH antagonist

INTERVENTIONS:
Drug: Growth hormone — Growth hormone is supplemented during the ovarian stimulation till the day of trigger
  Arms: GH group
Drug: GnRH antagonist — GnRH antagonist protocol for ovarian stimulation

SUMMARY:
This retrospective cohort study aims to investigate the effects of recombinant human growth hormone (rh-GH) on the euploid status of preimplantation blastocysts in AMA patients.

Infertile patients aged 38-46 years old were recruited for study if they fulfill the inclusion criteria and do not have the exclusion criteria.

Treatment group: Women received growth hormone (GH) supplement during antagonist protocol for ovarian stimulation.

Control group: Women received antagonist protocol for ovarian stimulation. The primary outcome is the euploidy rate of blastocysts per stimulation cycle and per testing cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age 38-46; BMI 18.5-24.0kg/m2; intended to undergo PGT-A; GnRH Antagonist protocol for ovarian stimulation; normal semen analysis for the male partner

Exclusion Criteria:

* Endometriosis grade 3 or higher, untreat hydrosalpinx;
* Women with a uterine cavity abnormality, such as a uterine congenital malformation (uterus uni-cornate, bicornate, or duplex);
* Untreated uterine septum, adenomyosis, submucous myoma, or endo-metrial polyp(s)
* Women who are indicated and planned to undergo PGT-SR (Preimplantation genetic testing for structural rearrangement) or PGT-M (Preimplantation genetic testing for monogenic disorder), for example, parental abnormal karyo-type or diagnosed with monogenic disease;
* Women who received other supplement drugs during ovarian stimulation

Ages: 38 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 692 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of cycles which obtained euploid blastocysts | 1 month after oocyte retrieval
  Number of cycles with at least 1 euploid blastocyst divided by the total number of stimulation cycles in a cohort

SECONDARY OUTCOMES:
Euploid blastocyst rate per cohort | 1 month after oocyte retrieval
  Total number of euploid blastocyst in a cohort/total number of biopsied embryos in the same cohort
Euploidy rate per cycle | 1 month after oocyte retrieval
  Euploidy rate of blastocysts, calculated per stimulation cycle and per testing cycle

OTHER OUTCOMES:
Embryo implantation | 14 days after embryo transfer
  Positive serum HCG 14 days after embryo transfer. Implantation rate=number of embryos implanted/embryo of embryos tranferred.
Clinical pregnancy | 30 days after embryo transfer
  Clinical pregnancy is defined as visualization of the gestational sac on ultrasonography. Clinical pregnancy rate=number of ongoing pregnancies/number of embryos transferred.
Ongoing pregnancy | 12 weeks' gestation
  Ongoing pregnancy is defined as a viable pregnancy beyond 12 weeks' gestation of the first frozen embryo transfer. Ongoing pregnancy rate=number of ongoing pregnancies/number of embryos transferred.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Sun, PhD, Study Director — Shanghai JIAI Genetics and IVF Institute
Locations (1):
- Shanghai JIAI Genetics and IVF Institute, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sui Y, Xiao M, Fu J, Li L, Xu Y, Lei C, Sun X. Growth hormone supplementation during ovarian stimulation in women with advanced maternal age undergoing preimplantation genetic testing for Aneuploidy. J Ovarian Res. 2023 Oct 19;16(1):204. doi: 10.1186/s13048-023-01279-y. PMID 37858247